CLINICAL TRIAL: NCT00727142
Title: Conservative Versus Surgical Management of Idiopathic Normal Pressure Hydrocephalus
Brief Title: Conservative Versus Surgical Management of Idiopathic Normal Pressure Hydrocephalus (INPH)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: observed benefit of treatment larger than expected
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, A Toma, Consultant Neurosurgeon, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08/0149
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: NPH; Hydrocephalus; Shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- open shunt (Active Comparator): functioning shunt
  Interventions: Procedure: Surgical treatment
- closed shunt (Active Comparator): NON FUNCTIONING SHUNT
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Insertion of a functioning shunt
  Other Names: Functioning shunt

SUMMARY:
This study aims to provide class 1 evidence supporting or refuting the existence of normal pressure hydrocephalus.

DETAILED DESCRIPTION:
By comparing one group with active CSF shunting with another with non .

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Normal pressure Hydrocephalus

Exclusion Criteria:

* Alzheimer disease
* Vascular dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
improvement in walking speed | 3 months

SECONDARY OUTCOMES:
improved cognition or continence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Watkins, FRCS, Principal Investigator — NHNN
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom